CLINICAL TRIAL: NCT05044481
Title: "Impact of the Third Molars in Oral Health-related Quality of Life"
Status: Completed | Type: Observational
Sponsor: Hospital Carlos Van Buren (Other)
Collaborators: Universidad de La Frontera (Other)
Responsible Party: Sponsor
Other Study IDs: ORD 1809 / 12-08-2019
Record Dates: First submitted 2021-09-12; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Health-related Quality of Life; Third Molar
Keywords: Health-related quality of life; third molar

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: third molar surgical removal — ambulatory surgical intervention of the maxilla and / or mandible for third molar removal

SUMMARY:
The aim of this study is to evaluate the impact of the third molars in oral health-related quality of life, before and after surgical removal using a validated and frequently used in international investigations instrument (OHIP-14).

DETAILED DESCRIPTION:
This is a prospective study that evaluates the oral health-related quality of life through the application of the self-administered OHIP-14 before and after the surgical removal of third molars. The inclusion criteria were adults' patients older than 18 years, referred for oral surgery. Patients with chronic diseases and acute pericoronitis were excluded. The assessment was performed at three times: pre-surgical planning 1 day before surgery (T0), 10 days (T1) and 2 - 3 months after surgery (T2)

ELIGIBILITY:
Inclusion Criteria:

* Adults patients over 18 years old

Exclusion Criteria:

* Patients with chronic diseases and acute pericoronitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old submmited to third molars surgical removal
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-06-14 (Actual)

PRIMARY OUTCOMES:
changes in oral health related quality of life after orthognathic surgery assessed with Short form Oral Health Impact Profile (OHIP-14) | baseline to 10 days and 2 - 3 months after surgery
  Short form Oral Health Impact Profile (OHIP-14) was applied at 3 times: baseline, one week before surgery (T1), 10 days after surgery (T2) and 2 - 3 months after surgery (T3).
  A paired t-test was used to assess the mean (SD) changes in patients undergoing orthognathic surgery. The magnitude of the change was evaluated calculating the standardized response mean (SRM).
  The Short Form Oral Health Impact Profile (OHIP-14) is an instrument for assessment oral health-related quality of life.
  14 ítems values: min = 0 / max = 56 higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Duarte, Principal Investigator — Hospital Carlos Van Buren
Locations (1):
- Valentina Duarte, Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No